CLINICAL TRIAL: NCT02558400
Title: A Prospective, Double-masked, Randomized, Multi-center, Active-controlled, Parallel-group 12-month Study Assessing the Safety and Ocular Hypotensive Efficacy of PG324 Ophthalmic Solution Compared to AR-13324 Ophthalmic Solution, 0.02% and Latanoprost Ophthalmic Solution, 0.005% in Subjects With Elevated Intraocular Pressure
Brief Title: Double-masked Study of PG324 Ophthalmic Solution in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PG324-CS301
Record Dates: First submitted 2015-09-16; First posted 2015-09-24 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — netarsudil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PG324 Ophthalmic Solution 0.02%/0.005% (Experimental): Fixed combination of netarsudil 0.02%, latanoprost 0.005% ophthalmic solution
  Interventions: Drug: PG324 Ophthalmic Solution 0.02%/0.005%
- AR-13324 Ophthalmic Solution 0.02% (Active Comparator): Netarsudil 0.02% ophthalmic solution
  Interventions: Drug: Netarsudil (AR-13324) Ophthalmic Solution 0.02%
- Latanoprost Ophthalmic Solution 0.005% (Active Comparator): Latanoprost 0.005% ophthalmic solution
  Interventions: Drug: Latanoprost Ophthalmic Solution 0.005%

INTERVENTIONS:
Drug: PG324 Ophthalmic Solution 0.02%/0.005% — 1 drop once daily (QD), in the evening (PM) in both eyes (OU)
  Arms: PG324 Ophthalmic Solution 0.02%/0.005%
Drug: Netarsudil (AR-13324) Ophthalmic Solution 0.02% — 1 drop once daily (QD), in the evening (PM) in both eyes (OU)
  Arms: AR-13324 Ophthalmic Solution 0.02%
Drug: Latanoprost Ophthalmic Solution 0.005% — 1 drop once daily (QD), in the evening (PM) in both eyes (OU)
  Arms: Latanoprost Ophthalmic Solution 0.005%

SUMMARY:
To evaluate ocular hypotensive efficacy and safety of PG324 Ophthalmic Solution compared to Netarsudil (AR-13324) Ophthalmic Solution and Latanoprost Ophthalmic Solution.

Following completion of the Month 12 study visit procedures, subjects will be offered the opportunity to participate in a 2-month observational (i.e., non-interventional) trial extension.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Diagnosis of open angle glaucoma or ocular hypertension in both eyes
3. Unmedicated intraocular pressure >20mmHg and <36mmHg in both eyes at 2 qualification visits. Both eyes had to qualify at all qualification visits
4. Corrected visual acuity equivalent to 20/200 Snellen or better
5. Able to give informed consent and follow study instructions

Exclusion Criteria:

1. Clinically significant ocular disease
2. Pseudoexfoliation or pigment dispersion component glaucoma, history of angle closure or narrow angles
3. Unmedicated Intraocular pressure ≥36mmHg
4. Use of more than 2 ocular hypotensive medications within 30 days of screening
5. Known hypersensitivity to any component of the formulation
6. Previous glaucoma surgery or refractive surgery
7. Ocular trauma within 6 months prior to screening
8. Any ocular surgery or non-refractive laser treatment within 3 months prior to screening
9. Recent or current ocular infection or inflammation in either eye
10. Used ocular medication in either eye of any kind within 30 days of screening
11. Mean central corneal thickness >620µm at screening
12. Any abnormality preventing reliable applanation tonometry of either eye
13. Clinically significant abnormalities in lab tests at screening
14. Clinically significant systemic disease
15. Participation in any investigational study within 60 days prior to screening
16. Used any systemic medication that could have a substantial effect on intraocular pressure within 30 days prior to screening
17. Women who are pregnant, nursing, planning a pregnancy or not using a medically acceptable form of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 718 (Actual)
Dates: Start 2015-09-18 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Heah, MD, MBA, Study Director — Aerie Pharmaceuticals, Inc.
Locations (1):
- Aerie Pharmaceuticals, Bedminster, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Asrani S, Bacharach J, Holland E, McKee H, Sheng H, Lewis RA, Kopczynski CC, Heah T. Fixed-Dose Combination of Netarsudil and Latanoprost in Ocular Hypertension and Open-Angle Glaucoma: Pooled Efficacy/Safety Analysis of Phase 3 MERCURY-1 and -2. Adv Ther. 2020 Apr;37(4):1620-1631. doi: 10.1007/s12325-020-01277-2. Epub 2020 Mar 12. PMID 32166538

RESULTS

PARTICIPANT FLOW:
Groups:
- PG324 Ophthalmic Solution 0.02%/0.005%: PG324 Ophthalmic Solution: 1 drop once daily (QD), in the evening (PM) in both eyes (OU)
Period: Overall Study
Arm/Group | PG324 Ophthalmic Solution 0.02%/0.005% | AR-13324 Ophthalmic Solution 0.02% | Latanoprost Ophthalmic Solution 0.005%
Started | 238 | 244 | 236
Completed | 159 | 148 | 203
Not Completed | 79 | 96 | 33
Not completed — Adverse Event | 47 | 53 | 4
Not completed — Withdrawal by Subject | 13 | 9 | 8
Not completed — Non-Compliant | 0 | 1 | 3
Not completed — Lost to Follow-up | 5 | 5 | 4
Not completed — Lack of Efficacy | 0 | 13 | 1
Not completed — Disallowed Concurrent Medication | 6 | 7 | 5
Not completed — Physician Decision | 2 | 2 | 0
Not completed — Protocol Violation | 6 | 3 | 8
Not completed — Death | 0 | 1 | 0
Not completed — Ineligible for the study | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- PG324 Ophthalmic Solution: PG324 Ophthalmic Solution: 1 drop once daily (QD), in the evening (PM) in both eyes (OU)
- Total: Total of all reporting groups
Arm/Group | PG324 Ophthalmic Solution | AR-13324 Ophthalmic Solution 0.02% | Latanoprost Ophthalmic Solution 0.005% | Total
Number analyzed (Participants) | 238 | 244 | 236 | 718
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 109 | 107 | 95 | 311
  >=65 years | 129 | 137 | 141 | 407
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (11.33) | 64.6 (10.97) | 65.4 (10.98) | 64.8 (11.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 136 | 136 | 406
  Male | 104 | 108 | 100 | 312
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 32 | 30 | 92
  Not Hispanic or Latino | 208 | 212 | 206 | 626
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 7 | 6 | 10 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 69 | 70 | 67 | 206
  White | 162 | 167 | 157 | 486
  More than one race | 0 | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: The primary efficacy variable was mean IOP at 08:00, 10:00 and 16:00 hours at Day 15, Day 43 and Day 90, as measured by Goldmann applanation tonometry. Secondary analysis were conducted as a part of safety measurements to month 12 on treatment.
Time Frame: Primary efficacy endpoint measured for 3 months (data collected at 08:00, 10:00 and 16:00 hours at Day 15, Day 43 and Day 90)
Population: Intent to Treat (ITT) population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PG324 Ophthalmic Solution | AR-13324 Ophthalmic Solution 0.02% | Latanoprost Ophthalmic Solution 0.005%
Number analyzed (Participants) | 238 | 244 | 236
mmHg
  Day 1, 0800 hours | 24.84 (3.316) | 24.81 (3.335) | 24.59 (2.914)
  Day 1, 1000 hours | 23.72 (3.587) | 23.45 (3.510) | 23.43 (3.385)
  Day 1, 1600 hours | 22.59 (3.610) | 22.63 (3.674) | 23.43 (3.370)
  Day 15, 0800 hours | 15.68 (3.532) | 18.66 (4.189) | 17.74 (3.467)
  Day 15, 1000 hours | 14.93 (3.417) | 17.78 (4.219) | 17.36 (3.548)
  Day 15, 1600 hours | 14.83 (2.978) | 17.25 (3.814) | 17.11 (3.236)
  Day 43, 0800 hours | 16.04 (3.268) | 19.06 (4.593) | 17.58 (3.465)
  Day 43, 1000 hours | 15.39 (3.175) | 17.92 (4.168) | 17.06 (3.250)
  Day 43, 1600 hours | 15.43 (3.065) | 17.54 (3.855) | 16.97 (3.240)
  Day 90, 0800 hours | 16.37 (3.377) | 19.04 (4.537) | 17.53 (3.280)
  Day 90, 1000 hours | 15.41 (3.038) | 17.96 (4.262) | 16.88 (3.139)
  Day 90, 1600 hours | 15.49 (3.126) | 17.30 (3.769) | 16.67 (3.115)
Statistical Analysis 1: Comparison: PG324 Ophthalmic Solution vs AR-13324 Ophthalmic Solution 0.02%; Test type: Superiority — To claim superiority PG324 had to be statistically superior to netarsudil and to latanoprost at all 9 of 9 primary efficacy timepoints; p < 0.0001, t-test, 2 sided; PG324 vs. netarsudil
Statistical Analysis 2: Comparison: PG324 Ophthalmic Solution vs Latanoprost Ophthalmic Solution 0.005%; Test type: Superiority; p < 0.0001, t-test, 2 sided; PG324 vs. latanoprost

2. Secondary Outcome: Extent of Exposure
Description: Exposure to study medication in days for all treatment groups
Time Frame: 12 months
Population: The safety population= all randomized subjects who received at least 1 dose of study medication. The safety population summarized subjects as-treated. 1 Subject was randomized to netarsudil but received latanoprost. Therefore, 1 less subject is in the netarsudil group and 1 additional subject is in the latanoprost group for the safety population.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PG324 Ophthalmic Solution 0.02%/0.005% | AR-13324 Ophthalmic Solution 0.02% | Latanoprost Ophthalmic Solution 0.005%
Number analyzed (Participants) | 238 | 243 | 237
days | 275.7 (129.94) | 266.2 (131.60) | 330.4 (89.60)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the course of the study of 12 month treatment and 2 month safety follow up.The safety population summarized subjects as-treated.
Description: Safety population, defined as all randomized subjects who received at least 1 dose of investigational product.The safety population summarized subjects as-treated. 1 Subject was randomized to netarsudil but received latanoprost. Therefore, 1 less subject is in the netarsudil group and 1 additional subject is in the latanoprost group for the safety population. (applies to the numbers of subjects for SAEs, all cause mortality and other AEs sections)
Arm/Group | PG324 Ophthalmic Solution | AR-13324 Ophthalmic Solution 0.02% | Latanoprost Ophthalmic Solution 0.005%
All-Cause Mortality (participants affected / at risk) | 0/238 | 1/243 | 0/237
Serious Adverse Events (participants affected / at risk) | 5/238 | 10/243 | 10/237
Other Adverse Events (participants affected / at risk) | 169/238 | 160/243 | 74/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PG324 Ophthalmic Solution (N=238) | AR-13324 Ophthalmic Solution 0.02% (N=243) | Latanoprost Ophthalmic Solution 0.005% (N=237)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastric Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Coronary Artery Stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PG324 Ophthalmic Solution (N=238) | AR-13324 Ophthalmic Solution 0.02% (N=243) | Latanoprost Ophthalmic Solution 0.005% (N=237)
Conjunctival Hyperaemia (Eye disorders) | 133 (133) | 115 (115) | 44 (44)
Cornea Verticillata (Eye disorders) | 39 (39) | 32 (32) | 0 (0)
Eye Pruritus (Eye disorders) | 20 (20) | 20 (20) | 2 (2)
Lacrimation Increased (Eye disorders) | 15 (15) | 17 (17) | 1 (1)
Conjunctival Haemorrhage (Eye disorders) | 10 (10) | 14 (14) | 2 (2)
Punctate Keratitis (Eye disorders) | 9 (9) | 13 (13) | 4 (4)
Vision Blurred (Eye disorders) | 9 (9) | 14 (14) | 3 (3)
Instillation Site Pain (General disorders) | 52 (52) | 55 (55) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT02558400/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT02558400/SAP_001.pdf